CLINICAL TRIAL: NCT02696772
Title: Effect of 24 h Severe Energy Restriction on Appetite Regulation and Ad-libitum Energy Intake in Lean Males and Females
Brief Title: Effect of 24 h Severe Energy Restriction on Appetite Regulation and Ad-libitum Energy Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loughborough University (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Lewis James, Lecturer in Nutrition, Loughborough University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: R13-P149DC
Record Dates: First submitted 2016-02-26; First posted 2016-03-02 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: Deficiency; Calorie
MeSH Terms: interventions — Energy Intake

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Energy balance (Experimental): Intervention day diet containing 100% of estimated energy requirements
  Interventions: Other: Energy intake
- Energy restriction (Experimental): Intervention day diet containing 25% of estimated energy requirements
  Interventions: Other: Energy intake

INTERVENTIONS:
Other: Energy intake

SUMMARY:
Long term maintenance of weight loss is generally poor, which is at least partly due to increased feelings of hunger associated with restricting what can be eaten. Intermittent severe energy restriction is a novel dietary strategy that requires individuals to consume a very-low energy diet for 1-4 days per week, allowing normal feeding patterns to be adopted on the other days in the week. However, the effect of a consuming a very-low energy diet on appetite regulation, which might represent a key marker of long-term adherence to dieting, has not been determined. This study aimed to assess the effects of severely restricting energy intake for 24 h on markers of appetite regulation, energy balance and metabolism compared to an adequate energy trial.

ELIGIBILITY:
Inclusion Criteria:

* non-smoker, not currently dieting, weight stable for >6 months (self-reported), no known history of cardiovascular or renal disease.

Exclusion Criteria:

* food allergies, dislike or intolerance of study foods and drinks, irregular eating patterns, use of medication that could influence hormone concentrations, excessive alcohol consumption (>4 units/day), intensive training schedule (>10 h/week)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2013-10; Primary Completion 2015-06 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Ad-libitum energy intake | 48 hours
  Measured at laboratory-based meals and weight food records
Subjective appetite | 48 hours
  Measured using visual analogue scales
Plasma acylated Ghrelin | 24 hours
  Measured using ELISA from venous blood samples
Plasma active glugagon-like peptide 1 | 24 hours
  Measured using ELISA from venous blood samples

SECONDARY OUTCOMES:
Plasma insulin | 24 hours
  Measured using ELISA from venous blood samples
Plasma glucose | 24 hours
  Measured using colorimetric assay from venous blood samples
Plasma Non-esterified Fatty acids | 24 hours
  Measured using colorimetric from venous blood samples
Energy expenditure | 24 hours
  Measured under resting conditions using indirect calorimetry
Fat oxidation | 24 hours
  Measured under resting conditions using indirect calorimetry
carbohydrate oxidation | 24 hors
  Measured under resting conditions using indirect calorimetry

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Clayton DJ, Burrell K, Mynott G, Creese M, Skidmore N, Stensel DJ, James LJ. Effect of 24-h severe energy restriction on appetite regulation and ad libitum energy intake in lean men and women. Am J Clin Nutr. 2016 Dec;104(6):1545-1553. doi: 10.3945/ajcn.116.136937. Epub 2016 Nov 2. PMID 27806971